CLINICAL TRIAL: NCT05869903
Title: A Phase 3, Randomized, Double-Blind Study to Investigate the Efficacy and Safety of Once-Daily Oral Orforglipron Compared With Placebo in Adult Participants With Obesity or Overweight With Weight-Related Comorbidities (ATTAIN-1)
Brief Title: A Study of Orforglipron (LY3502970) in Adult Participants With Obesity or Overweight With Weight-Related Comorbidities
Acronym: ATTAIN-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18559; J2A-MC-GZGP (Other: Eli Lilly and Company); 2022-502839-19-00 (Other: Eli Lilly and Company); U1111-1289-8877 (Other: UTN Number)
Record Dates: First submitted 2023-05-12; First posted 2023-05-22 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Overweight; Overweight or Obesity
MeSH Terms: conditions — Obesity; Overweight | interventions — orforglipron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Orforglipron Dose 1 (Experimental): Participants will receive orforglipron administered orally.
  Interventions: Drug: Orforglipron
- Orforglipron Dose 2 (Experimental): Participants will receive orforglipron administered orally.
  Interventions: Drug: Orforglipron
- Orforglipron Dose 3 (Experimental): Participants will receive orforglipron administered orally.
  Interventions: Drug: Orforglipron
- Placebo (Placebo Comparator): Participants will be given placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orforglipron — Administered orally.
  Other Names: LY3502970
  Arms: Orforglipron Dose 1; Orforglipron Dose 2; Orforglipron Dose 3
Drug: Placebo — Administered orally.
  Arms: Placebo

SUMMARY:
This study will investigate the efficacy and safety of once daily oral orforglipron in adult participants with obesity or overweight with weight-related comorbidities. The study has two phases: a main phase and an extension phase. The main phase of the study lasted 72 weeks. Participants with prediabetes will continue in the extension for another 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Have a BMI

  * ≥30.0 kilogram/square meter (kg/m²),
  * ≥27.0 kg/m² and presence of at least 1 of the following weight-related comorbidities (treated or untreated) at screening:

    * Hypertension, dyslipidemia, obstructive sleep apnea, cardiovascular disease (for example, ischemic cardiovascular disease, New York Heart Association Functional Class I-III heart failure).
* Have a history of at least 1 self-reported unsuccessful dietary effort to lose body weight.

Exclusion Criteria:

* Have Type 1 diabetes, Type 2 diabetes, or any other types of diabetes, history of ketoacidosis, or hyperosmolar state/coma
* Have a self-reported change in body weight >5 kg (11 pounds) within 90 days prior to screening.
* Have family (first-degree relative) or personal history of medullary thyroid cancer (MTC) or multiple endocrine neoplasia (MEN)2 syndrome.
* Have had a history of chronic or acute pancreatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3127 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Mean Percent Change from Baseline in Body Weight | Baseline to Week 72

SECONDARY OUTCOMES:
Mean Change from Baseline in Waist Circumference | Baseline, Week 72
Mean Change from Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 72
Mean Percent Change from Baseline in Fasting non-HDL Cholesterol | Baseline, Week 72
Mean Percent Change from Baseline in Fasting Triglycerides | Baseline, Week 72
Mean Change from Baseline in Hemoglobin A1c (HbA1c) % | Baseline, Week 72
Mean Change from Baseline in Fasting Glucose | Baseline, Week 72
Mean Percent Change from Baseline in Fasting Insulin | Baseline, Week 72
Mean Change from Baseline in Diastolic Blood Pressure (DBP) | Baseline, Week 72
Mean Change from Baseline in Short Form Version 2 (SF-36v2) Acute Form Domain Scores | Baseline, Week 72
Mean Percent Change from Baseline in Body Weight in Participants with Prediabetes at Randomization | Baseline, Week 176
Time to Onset of Type 2 Diabetes | Baseline through Week 176, Baseline through Week 190

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (138):
- United States (43):
  - The Institute for Liver Health II dba Arizona Clinical Trials - Mesa, Chandler, Arizona
  - Clinical Research Institute of Arizona (CRI) - Sun City West, Sun City West, Arizona
  - John Muir Physician Network Research Center, Concord, California
  - AMCR Institute, Escondido, California
  - NorCal Medical Research, Inc, Greenbrae, California
  - Velocity Clinical Research, Huntington Park, Huntington Park, California
  - Velocity Clinical Research, Westlake, Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - Norcal Endocrinology & Internal Medicine, San Ramon, California
  - University Clinical Investigators, Inc., Tustin, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - New Age Medical Research Corporation, Miami, Florida
  - South Broward Research, Miramar, Florida
  - Renstar Medical Research, Ocala, Florida
  - Jedidiah Clinical Research - Tampa - Bay Plaza, Tampa, Florida
  - Clinical Site Partners, LLC dba Flourish Research, Winter Park, Florida
  - Physicians Research Associates, Lawrenceville, Georgia
  - East Coast Institute for Research, LLC, Macon, Georgia
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Elite Clinical Trials, Blackfoot, Idaho
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Cotton O'Neil Diabetes & Endocrinology, Topeka, Kansas
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Care Access - Lake Charles, Lake Charles, Louisiana
  - MedStar Health Research Institute (MedStar Physician Based Research Network), Hyattsville, Maryland
  - Endocrine and Metabolic Consultants, Rockville, Maryland
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - SKY Integrative Medical Center/SKYCRNG, Ridgeland, Mississippi
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Long Island Cardiovascular Consultants, Lake Success, New York
  - Weill Cornell Medical College, New York, New York
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Thyroid, Endocrinology, and Diabetes, Dallas, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - Cedar Health Research, Dallas, Texas
  - Juno Research, Houston, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Soma Clinical Trials, Wylie, Texas
  - Physicians' Research Options, Draper, Utah
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - Eastside Research Associates, Redmond, Washington
- Brazil (14):
  - Centro de Pesquisas em Diabetes e Doenças Endócrino-Metabólicas, Fortaleza, Ceará
  - CEDOES, Vitória, Espírito Santo
  - Hospital São Domingos, Bequimão, Maranhão
  - Cline Research Center, Curitiba, Paraná
  - Quanta Diagnóstico e Terapia, Curitiba, Paraná
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Sao Lucas, Campinas, São Paulo
  - CECIP - Centro de Estudos do Interior Paulista, Jaú, São Paulo
  - Centro Multidisciplinar de Estudos Clinicos, São Bernardo do Campo, São Paulo
  - Integral Pesquisa e Ensino, Votuporanga, São Paulo
  - Hospital São Lucas de Copacabana, Rio de Janeiro
  - CPQuali Pesquisa Clínica, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
  - Hospital das Clinicas FMUSP, São Paulo
- China (20):
  - The Second People's Hospital of Hefei, Hefei, Anhui
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Chongqing General Hospital, Chongqing, Chongqing Municipality
  - ShenZhen People's Hospital, Shenzhen, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Jinan Central Hospital, Jinan, Shandong
  - Jiading District Central Hospital, Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Zhu Xianyi Memorial Hospital, Tianjin, Tianjin Municipality
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
- India (8):
  - Endolife Speciality Hospitals, Guntur, Andhra Pradesh
  - Victoria Hospital, Bangalore Medical College And Research Institute, Bangalore, Karnataka
  - Mysore Medical College, Mysore, Karnataka
  - Central India Cardiology and Research Institute, Nagpur, Maharashtra
  - All India Institute of Medical Sciences (AIIMS) - Nagpur, Nagpur, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - Lifepoint Multispeciality Hospital, Pune, Maharashtra
- Japan (18):
  - Oishi Clinic, Wakasugi, Fukuoka
  - Mazda Hospital, Aki-gun, Hiroshima
  - Tsuchiura Medical & Health Care Center, Tsuchiura, Ibaraki
  - NTT Nishinihon Takamatsu Clinic, Takamatsu, Kagawa-ken
  - Iwamoto Internal Medicine Clinic, Zentsujichó, Kagawa-ken
  - Yokohama Minoru Clinic, Yokohama, Kanagawa
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi, Osaka
  - Sugiura Internal Medicine Clinic, Sōka, Saitama
  - Adachi Kyosai Hospital, Adachi-ku, Tokyo
  - Medical Corporation Chiseikai Tokyo Center Clinic, Chuo-ku, Tokyo
  - Tokyo-Eki Center-building Clinic, Chuo-ku, Tokyo
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Yutenji Medical Clinic, Meguro-ku, Tokyo
  - Kanno Naika, Mitaka, Tokyo
  - Shimokitazawa Tomo Clinic, Setagaya-ku, Tokyo
  - Heishinkai Medical Group ToCROM Clinic, Shinjuku-ku, Tokyo
  - Boocs Clinic Fukuoka, Fukuoka
  - Osaka Nishiumeda Clinic, Osaka
- Puerto Rico (2):
  - GCM Medical Group, PSC - Hato Rey Site, San Juan, PR
  - Dorado Medical Complex, Dorado
- Slovakia (8):
  - Nemocnica s poliklinikou Lucenec, Lučenec, Banská Bystrica Region
  - Metabol KLINIK, Bratislava, Bratislava Region
  - Human Care s.r.o., Košice, Košice Region
  - Areteus s.r.o., Trebišov, Košice Region
  - DIAB sro, Rožňava, Košický Kr
  - MEDI-DIA s.r.o., Sabinov, Presov
  - DIA-MED CENTRUM s.r.o., Púchov, Trenčín Region
  - MediTask, Bratislava
- South Korea (7):
  - Gachon University Gil Medical Center, Namdong-gu, Incheon-gw
  - Korea University Ansan Hospital, Ansan-si, Kyǒnggi-do
  - Hallym University Sacred Heart Hospital, Anyang-si, Kyǒnggi-do
  - Ajou University Hospital, Suwon, Kyǒnggi-do
  - Pusan National University Yangsan Hospital, Busan, Kyǒngsangnam-do
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Konyang University Hospital, Seogu, Taejǒn-Kwangyǒkshi
- Spain (13):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña [La Coruña]
  - Complejo Hospitalario Universitario de Ferrol (CHUF)- Hospital Naval, Ferrol, A Coruña [La Coruña]
  - Centro Periférico de Especialidades Bola Azul, Almería, Almería
  - Hospital Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Quiron Infanta Luisa, Seville, Andalusia
  - Hospital Germans Trias i Pujol, Badalona, Barcelona [Barcelona]
  - Centro Médico Teknon, Barcelona, Barcelona [Barcelona]
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Hospital Clínico Universitario de Valladolid, Valladolid, Castille and León
  - Hospital Virgen del Camino, Sanlúcar de Barrameda, Cádiz
  - Hospital Virgen de las Montañas, Villamartín, Cádiz
  - Hospital General Universitario de Valencia, Valencia, Valenciana, Comunitat
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (5):
  - Chiayi Christian Hospital, Chiayi City, Chiayi
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist, Kaohsiung
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Wharton S, Aronne LJ, Stefanski A, Alfaris NF, Ciudin A, Yokote K, Halpern B, Shukla AP, Zhou C, Macpherson L, Allen SE, Ahmad NN, Klise SR; ATTAIN-1 Trial Investigators. Orforglipron, an Oral Small-Molecule GLP-1 Receptor Agonist for Obesity Treatment. N Engl J Med. 2025 Nov 6;393(18):1796-1806. doi: 10.1056/NEJMoa2511774. Epub 2025 Sep 16. PMID 40960239
- See also: A Study of Orforglipron (LY3502970) in Adult Participants With Obesity or Overweight With Weight-Related Comorbidities (ATTAIN-1) — https://trials.lilly.com/en-US/trial/403875